CLINICAL TRIAL: NCT06153173
Title: A Phase II Trial of the MEK Inhibitor Mirdametinib in Histiocytic Disorders
Brief Title: Mirdametinib in Histiocytic Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0206
Record Dates: First submitted 2023-10-11; First posted 2023-12-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Langerhans Cell Histiocytosis (LCH); Juvenile Xanthogranuloma (JXG); Rosai-Dorfman Disease (RDD); Histiocytic Disorders
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Xanthogranuloma, Juvenile; Histiocytosis, Sinus | interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirdametinib (Experimental): Mirdametinib will be dosed by mouth twice a day at a dose of 2 mg/m2 BID with a max of 4 mg BID (8 mg per day max).
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Mirdametinib — Mirdametinib is administered by mouth twice daily on a continuous schedule, with each cycle being 4 weeks. Patients are instructed to take consecutive doses separated by a minimum of 6 hours and a maximum of 14 hours.

SUMMARY:
The purpose of this study is to see if treatment with mirdametinib in patients with Langerhans cell histiocytosis (LCH) or other histiocytic disorders will be better than current treatments and with fewer side effects.

DETAILED DESCRIPTION:
Langerhans cell histiocytosis (LCH) is a rare blood disorder. Though affecting all ages, LCH occurs more often in children, with an increased incidence in children less than 1 year of age. The disease presents in various ways, with most children suffering bony lesions, and skin rashes. In some patients, LCH affects vital organs such as liver, spleen, bone marrow, and the central nervous system. This group of patients are at significant risk of serious illness and death and are thus said to have risk-organ-positive (RO+) LCH. Current treatments for LCH consist of chemotherapy combined with other medications. However, many patients, especially those with RO+ disease, do not respond to therapy. Of the patients that do respond, many suffer progression of disease after an initial response to therapy, or recurrence of disease after completion of therapy.

The purpose of this study is to see if treatment with mirdametinib in patients with LCH or other histiocytic disorders will be better than current treatments and with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥ 2 years of age AND have a diagnosis of a histiocytic disorder that requires systemic therapy

   * If patient has had a diagnostic biopsy, biopsy must be reviewed and confirmed by CCHMC pathologist as feasible
   * If patient has had a biopsy but has not had molecular testing done, must have tissue available for mutational analysis
   * If patient has isolated pituitary/CNS disease or situations where biopsy is not feasible, positive ddPCR blood test for mutation associated with histiocytic neoplasm with clinical features of histiocytosis is sufficient
2. Must have measurable disease on PET scan or brain MRI
3. Subjects must demonstrate adequate organ function as defined:

   * Renal: maximum serum creatinine 2x the upper limit of normal (ULN) OR a creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2
   * Liver: ALT ≤ 3x ULN AND normal INR (≤ 1.5)
   * Hematologic: Hematology: Albumin ≥ 2.8 g/dL; Absolute neutrophil count ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hemoglobin ≥ 9.0 g/dL
   * Patients with organ function abnormalities outside of these thresholds deemed to be the result of histiocytic disease will be considered eligible

Exclusion Criteria:

1. Prior therapy with stipulations as described:

   * Myelosuppressive Chemotherapy: Must not have received any cytotoxic chemotherapy which impacts the growth and development of cells in the bone marrow within 14 days of enrollment onto this study (i.e. cytarabine, cladribine, clofarabine, mercaptopurine, methotrexate, vinblastine)
   * MEK Inhibitors: Must not have received a MEK inhibitor within 30 days (or 5 half-lives, whichever is longer) of enrollment, NOR have had disease progression on MEK inhibitor
   * Steroids: Due to the increased risk of an ocular event, the use of systemic oral, inhaled, or ocular glucocorticoid therapy is prohibited within 14 days prior to first dose of mirdametinib. Throughout the treatment period, short term glucocorticoid treatment (30 days or less) is permitted. Any patients requiring long-term steroid use (more than 30 consecutive days) are not eligible. The exception to this rule is subjects with endocrine deficiencies who require physiologic steroids
   * Radiation: Must not have received radiation within 14 days of study enrollment or have received radiation to the orbit at any time
2. Risk factors for retinal vein occlusion (RVO) are listed. Exclusion should be considered by clinical discretion if they have any of the following risk factors for RVO at screening:

   * Intraocular pressure (IOP) > 21 mmHg; if IOP is unable to be obtained (eg age, cooperation, tolerability), ophthalmologist's exam findings and overall assessment will be utilized. If in the ophthalmologist's assessment there are no signs of raised IOP, the subject will be considered eligible for this parameter
   * Glaucoma or any significant abnormality (≥ grade 2) on ophthalmologic exam that is uncontrolled with intervention
   * Serum cholesterol > 300 mg/dL
   * Serum triglycerides > 300 mg/dL
   * Hyperglycemia (either fasting blood glucose > 125 mg/dL OR random blood glucose > 200 mg/dL)
   * Uncontrolled hypertension (participants ≤ 12 years of age with a blood pressure ≥ 95th percentile for age + 12 mmHg; participants ≥ 13 years of age with a blood pressure ≥ 140/90 mm Hg) unresolved on repeat measurement
3. LVEF < 55% at screening OR history of clinically significant cardiac disease, unless deemed to be the direct result of disease
4. Subjects who are pregnant or breastfeeding, or are at risk of pregnancy or fathering a baby and are unable to use acceptable methods of birth control during the length of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Response rate to mirdametinib | 1 year (completion of 13 four week cycles)
  Best overall response rate to mirdametinib after 13 four-week cycles as defined by positron emission tomography (PET) or magnetic resonance imaging (MRI) (for isolated pituitary/central nervous system (CNS) disease) response criteria.

SECONDARY OUTCOMES:
Duration of response to mirdametinib | 2 years (completion of 26 four week cycles)
  Duration of response to mirdametinib on study as defined by PET or MRI (for isolated pituitary/CNS disease) response criteria.
Maximum Plasma Concentration (Cmax) | Day 1 of the first 5 four week cycles)
  Blood samples will be drawn for the pharmacokinetic profile before, and during mirdametinib therapy. Maximum plasma concentration will be calculated as data allow.
Time to peak drug concentration (Tmax) | Day 1 of the first 5 four week cycles)
  Blood samples will be drawn for the pharmacokinetic profile before, and during mirdametinib therapy. Time to peak drug concentration (Tmax) will be calculated as data allow.
Area under the plasma concentration time curve (AUC) | Day 1 of the first 5 four week cycles)
  Blood samples will be drawn for the pharmacokinetic profile before, and during mirdametinib therapy. Area under the plasma concentration time curve (AUC) will be calculated as data allow.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Kumar, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Allison Bartlett, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States